CLINICAL TRIAL: NCT01837381
Title: A Comprehensive Analysis of Clinical Outcome, Treatment Toxicity and Tumor Response of Transarterial Ablation(TEA) for Unresectable Hepatocellular Carcinoma(HCC)
Brief Title: Transarterial Ethanol Ablation(TEA) for Unresectable Hepatocellular Carcinoma(HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-13-03
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transarterial Ethanol Ablation (TEA) (Other): Two treatment sessions at 2 months apart were given and started within 4 weeks after randomization.
  Interventions: Procedure: TEA

INTERVENTIONS:
Procedure: TEA — Arterial feeders to tumors were identified and catheterized with a microcatheter to a branch supplying a Couinaud segment or subsegmental level for delivery of the therapeutic agent, which was Lipiodol-ethanol mixture at 2:1 ratio by volume for TEA (Lipiodol Ultrafluide, Guerbet, France; Dehydrated alcohol [absolute alcohol], Martindale Pharmaceuticals, United Kingdom). The agents were delivered under fluoroscopic control to completely fill up the vasculature of all tumors. The maximum total volume of Lipiodol-ethanol mixture or cisplatin emulsion to be delivered in one treatment session was 60 mL.

SUMMARY:
The objective of this trial was to evaluate the clinical outcome, treatment toxicity and tumor response of TEA for unresectable HCC.

DETAILED DESCRIPTION:
Transarterial therapy has been playing an important role in the treatment algorithm for patients with multifocal or large intrahepatic lesions not eligible for surgical resection, transplantation, or local ablative therapy. Among the various options of transarterial therapy including chemoembolization (TACE), bland embolization, radioembolization, and TEA, chemoembolization is the only one that has been proven to be of survival benefits versus best supportive care in randomized controlled trials. TEA is a hybrid of bland embolization and chemical ablation. Utilizing a liquid agent of Lipiodol-ethanol mixture consisting of 33% ethanol by volume, TEA offers complete and long lasting embolization of both the arterioles and portal venules supplying the tumor and could possibly be more effective than particulate embolic agents in tumor vessel embolization. The component of ethanol very likely offers synergistic effect to embolization and causes tumor ablation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by patient
* Age above 18 years
* Child-Pugh A or B cirrhosis
* Eastern Cooperative Oncology Group(ECOG) performance score 2 or below
* No serious concurrent medical illness
* No prior treatment or surgery for HCC
* Histologically or cytologically proven HCC except for lesions of size 1 to 2 cm, with typical features of HCC on two dynamic imaging techniques, or lesions larger than 2cm, with typical features on one dynamic imaging techniques, or lesions larger than 2cm with alpha feto protein(AFP) level > 200 ng/mL
* Unresectable disease without extra-hepatic involvement on chest X-ray(CXR) and CT
* Massive expansive tumor type with measurable lesion on CT
* Total tumor mass < 50% liver volume
* Tumor size ≤ 15cm in largest dimension
* Tumor number ≤ 5

Exclusion Criteria:

* History of prior malignancy except on the condition that the patient has been disease free for ≥ 3 years
* Concurrent ischemic heart disease or heart failure
* History of acute tumor rupture presenting with hemo-peritoneum
* Serum creatinine level > 180 umol/L
* Biliary obstruction not amenable to percutaneous drainage
* Child-Pugh C cirrhosis
* History of hepatic encephalopathy
* Intractable ascites not controllable by medical therapy
* History of variceal bleeding within last 3 months; serum total bilirubin level ≥ 50 umol/L
* Serum albumin level < 25g/L
* International normalized ratio(INR) > 1.5
* Extrahepatic metastasis
* Infiltrative or diffuse tumor
* Tumor number > 5
* Thrombosis of target hepatic artery
* Partial or complete thrombosis of the main portal vein; tumor invasion of portal branch of contralateral lobe
* Hepatic vein tumor thrombus
* Significant arterio-portal venous shunt
* Significant arterial-hepatic venous shunt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
overall survival and treatment-related toxicity | Overall survival is studied from treatment to death from any cause, for an estimated period of up to 60 months. Treatment-related toxicity is studied up to 3 months after treatment
  Overall survival was defined as date of treatment to date of death from any cause. Patients alive at the end of follow-up were censored.
  Clinical and laboratory data were documented prospectively at baseline, during hospitalization, and at 7, 14, and 30 day, and 3, 6, 9, and 12 months. Laboratory findings were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.

SECONDARY OUTCOMES:
Time to progression(TTP) | Time to progression is studied from treatment to disease progression, for an estimated period of up to 60 months.
  TTP was defined as date of treatment to date of first CT evidence of disease progression. Patient death during follow-up without CT progression was censored.
Progression free survival(PFS) | Progression free survival is studied from treatment to disease progression or death from any cause, for an estimated period of up to 60 months.
  PFS was defined as date of treatment to date of either first CT evidence of disease progression or death from any cause. Patients alive and free of progression at the end of follow-up were censored.
Tumor response | Tumor response is studied at 6 months after treatment
  Treatment response of individual treated tumor lesions was evaluated with CT and classified according to a system combining the recommendation of European Association for the Study of the Liver and the guidelines of World Health Organization, which was considered a preferred method of response assessment following transarterial or locoregional therapies for HCC. Tumor response was classified into 4 categories: 1) complete response (CR), 2) partial response (PR), 3) static disease (SD), or 4) intralesional progression.

CONTACTS AND LOCATIONS:
Overall Officials: Simon CH Yu, MD, FRCR, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Department of Clinicl Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinsese University of Hong Kong, Hong Kong
  - Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No